CLINICAL TRIAL: NCT07286669
Title: Positional Release Technique of Iliotibial Band and Pes Anserine Versus Proprioception Exercise on Patients With Knee Osteoarthritis
Acronym: PRT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nabil Mahmoud Ismail Abdel-Aal, principle investigator : nabil mahmoud ismail, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/006112
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Positional Release Technique; Proprioception Exercise; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: positional release technique and proprioception exrecises
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Positional Release Technique (Experimental): Twenty patients will receive positional release technique in addition to traditional exercises. The treatment protocol will be 3 sessions per week for six weeks
  Interventions: Other: Positional Release Technique; Other: traditional exercise
- proprioception exercises (Experimental): Twenty patients will receive proprioception exercises in addition to traditional exercise. The treatment protocol will be 3 sessions per week for six weeks.
  Interventions: Other: proprioception exercises; Other: traditional exercise
- traditional exercise (Active Comparator): Twenty patients receive only traditional exercise. Treatment protocol will be 3 session per week for six weeks
  Interventions: Other: traditional exercise

INTERVENTIONS:
Other: Positional Release Technique — Positional release of Pes Anserine:Slide the fingers approximately 1 inch (2.5 cm) medially from the tibial tuberosity onto the bony insertion site. On the well-developed patient, the mass of the tendons can be grasped as a group at the medial knee.Apply tibial traction or upward compression with the far hand for fine-tuning. Maintain for 90 seconds with repeation 3 times in a session with a break of 30 seconds. Positional release of iliotibial band:Stand on the side of the supine patient that is opposite the band to be palpated. With your hands flat, align them over the lateral thigh just below the greater trochanter of the femur.
  Apply cephalad compression of the limb with the far hand or your body to fine-tune. Maintain for 90 seconds with repetition 3 times in a session with a break of 30 seconds
  Arms: Positional Release Technique
Other: proprioception exercises — the patients will receive proprioceptive exercises in the form of Heel Walk, Toe Walk, Sideways Knitting Walk, Sideways Step,Cross Walk, Semi Tandem Walk, Tandem Walk, High Knee Walk, Wedding Walk, Backward Wedding Walk, balance and coordination exercises.
  Arms: proprioception exercises
Other: traditional exercise — Stretch exercises: Rectus femoris, Iliotibial band, Hamstring and stretch for calf muscle (3sets, each stretch 30 sec hold, 30 second relaxation between each set 5sec rests). and repeated 3 times.
  Strengthen exercises: Isometric Exercises for quadriceps (10 rep,3sets), Hip abductors strengthening 45 degree (10 rep,3sets), Hip extensor strengthening 15 degree (10 rep,3sets), Straight leg raising 45-70 degree (10 rep,3sets), Short arc knee extension (10 rep,3sets)

SUMMARY:
this studty was conducted to compare the effect of the positional release technique of the iliotibial band and Pes Anserine Versus Proprioception Exercise on Patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is one of the most common chronic diseases in the world. It is frequently accompanied by high levels of persistent pain. Osteoarthritis is the most common degenerative disease, primarily affects the articular cartilage and the subchondral bone of a synovial joint, eventually resulting in joint failure. It is a disease involving multiple alterations on the joint tissues, including cartilage degradation, bone remodeling, and osteophyte formation; this leads to clinical manifestations, including pain, stiffness, swelling, and limitations in joint function. The positional release technique is a type of manual therapy that can be used effectively in treating pain and disability that is associated with musculoskeletal dysfunctional conditions and decrease tissue tenderness by altering nociceptor activity in the soft tissues. The positional release appears to affect inappropriate proprioceptive activity, thus helping to normalize tone and set the normal length-tension relationship in the muscle. Proprioceptive exercise is an effective way to strengthen knee joint muscle function and reduce pain in patients with knee osteoarthritis. The current study, it may be useful to compare the effect of the positional release technique, as it is a new modality and has proven its effectiveness in several studies on decreasing pain and dysfunction and increasing range of motion, versus the proprioception exercises which also have an improvement on pain, range, and function. The knee proprioception and pain pressure threshold will be also tested to compare these techniques on knee osteoarthritis patients

ELIGIBILITY:
Inclusion Criteria:

* Both genders with knee osteoarthritis will participate in this study according to the American College of Rheumatology criteria
* An average pain intensity of ≥3 on a 10-cm visual analogue scale (VAS).
* Patients with unilateral knee osteoarthritis, for those patients with bilateral knee -Patients with grade II &lll chronic knee osteoarthritis (clinical and imaging diagnosis X-ray.
* Patients were referred by orthopedic physician.
* Patients with body mass index <30Kg/cm2.

Exclusion Criteria:

* Previous knee surgery
* Serious valgus or varus deformity
* Past or present vascular disorder.
* Acute or chronic low back pain.
* Upper motor neuron lesion and lower motor neuron lesion.
* A history of rheumatoid arthritis.
* Presence of malignancy.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
knee disabiity | up to 6 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) was widely used in the evaluation of Hip and Knee Osteoarthritis. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales;Pain (5 items),Stiffness (2 items), Physical Function (17 items): The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations

SECONDARY OUTCOMES:
pain intensity | up to 6 weeks
  Patients recorded pain intensity on a 100 mm VAS by drawing a vertical line on the horizontally positioned VAS. The left end of the VAS represented 'no pain' and the right end 'most severe pain imaginable' with no intermediate divisions or descriptive terms
range of motion | up to six weeks
  The most often used clinical instrument for assessing joint AROM is the digital goniometer. It is used as a valid and reliable AROM measurement device with a high validity, intra- rater and inter-rater reliability
pressure pain threshold | up to six weeks
  The pressure algometer will be used to measure pressure pain threshold
knee joint position error | up to six weeks
  Free inclinometer application (Goniometer Pro, 5fuf5, USA) for iPhone 6 (Apple, Cupertino, USA) at 30°, 45° and 75° target angles. Active knee joint position sense will be assessing by iPhone inclinometer application. All tests will be performed at sitting position without any contact of the feet to the floor, at a quiet place and with closed eyes